CLINICAL TRIAL: NCT01927679
Title: Effect of Vitamin E in the Prevention of Visible Light Induced Pigmentation
Brief Title: Vitamin E Prevention of Visible Light Pigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Inno-6031
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Pigmentation From Visible Light
MeSH Terms: interventions — Vitamin E; Antioxidants; eucerin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antioxidant (LB) + control (UB) (Other): Antioxidant will be weighed and applied to an area on the lower back (LB) to be exposed with visible light at a concentration of 2 mg/cm^2. Control will also be weighed and applied to an area of the upper back (UB) to be exposed with visible light at a concentration of 2 mg/cm^2. These will be applied according to the randomization scheme.
  Interventions: Drug: Vitamin E; Drug: Eucerin
- Antioxidant (UB) and Control (LB) (Other): Antioxidant will be weighed and applied to an area on the upper back (UB) to be exposed with visible light at a concentration of 2 mg/cm^2. Control will also be weighed and applied to an area of the lower back (LB) to be exposed with visible light at a concentration of 2 mg/cm^2. These will be applied according to the randomization scheme.
  Interventions: Drug: Vitamin E; Drug: Eucerin

INTERVENTIONS:
Drug: Vitamin E
  Other Names: Antioxidant
Drug: Eucerin — Control

SUMMARY:
The main objective of the study is to assess the efficacy of an antioxidant in preventing pigmentation induced by visible light in subjects with a phototype IV or V.

Patients will be exposed to a range of visible light to areas on the back to confirm study eligibility. Patients showing pigmentation after 7 days on the exposed areas will be eligible to continue.

Eligible patients will have study product applied to part of the back and placebo on another part of the back. The placebo area will be exposed to the same range of light based as at Day -7. The area where the antioxidant is applied will have a higher range of light exposure than the area without the study product.

Seven days later, the areas will be examined to determine the lowest exposure inducing pigmentation on the sides with placebo and with antioxidant. The color will also be measured between two identical exposures with placebo and with antioxidant.

DETAILED DESCRIPTION:
At Day -7, all subjects will be exposed to a pre-specified range of doses of visible light on 6 areas of the back, each measuring 0.9 cm^2 in order to evaluate their pigmentary response to visible light. The doses will be 20, 40, 80, 160, 320 and 640 J/cm^2. At Day 0, a visual inspection will establish which subjects qualify for the remainder of the study, based on the presence or absence of pigmentation induced by visible light. Subjects who do not exhibit pigmentation at 640 J/cm^2 or lower will not pursue the study.

Subjects who demonstrate pigmentation will move on to the next step of the study. On this same Day 0 visit, these subjects will be randomized to receive a topical antioxidant preparation on one of two halves of their back and a control on the other side. The antioxidant and control will be applied twice before the exposure to visible light is done on Day 1: 24 hours prior (Day 0) and 30 minutes prior (Day 1) exposure. On Day 1, the skin with antioxidant will be exposed to fluences of 80, 160, 320, 640, 1280 and 1920 J/cm^2 whereas that with control will be exposed to the same lower doses as on Day -7. This will be done on a total of 12 different areas of 0.9 cm^2 each, with six on the side with antioxidant preparation, and six on the side with control.

On Day 7±1, a visual assessment will be done of each exposed area, as well as quantitative colorimetric measurements and a research photograph. The visual assessment will consist in determination of the lowest fluence inducing visible pigmentation on each half back (with antioxidant and with control). The colorimetric measurements will be done on areas exposed to 320 and 640 J/cm^2 to compare the pigmentation present on skin to which antioxidant was applied and on skin to which control was applied. The colorimetric assessment of adjacent unexposed skin will also be performed. At Day 0, 1 and 7 visits, subjects will also be evaluated for adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18 years of age or older at time of consent.
2. Subject, male or female, is willing to use effective contraceptive method for at least 30 days before Day -7 and at least until Day 7±1. Effective contraceptive methods are:

   1. Barrier methods such as condom, sponge or diaphragm combined with spermicide in foam, gel or cream;
   2. Hormonal contraception (oral, intramuscular, implant or transdermal) which include Depo-Provera, Evra and Nuvaring;
   3. Intrauterine device (IUD);
   4. Sterilization such as tubal ligation, hysterectomy or vasectomy;
   5. Postmenopausal state for at least 1 year for female subject or female partner of male subject;
   6. Same-sex partner;
   7. Abstinence.
3. Capable of giving informed consent and the consent must be obtained prior to any study related procedures.
4. Skin phototype IV and V
5. Exhibits visible light-induced pigmentation at Day 0
6. Is willing to avoid exposure to UV radiation, including sunlight, phototherapy, or tanning salon, on the back for the duration of the study and 4 weeks preceding the study.

Exclusion Criteria:

1. Current pregnancy or lactation
2. Allergy to any of the products used in the study
3. Use of phototherapy or tanning beds within the 30 days of the study start (Day -7)
4. Use of photosensitizing medication within the 30 days or 5 half-lives (whichever is longest) from the study start (Day-7)
5. Use of products other than the ones used in the study that may alter the pigmentation of the skin
6. Skin condition or medical condition altering the appearance of the skin in the area to be irradiated that would interfere with pigmentation evaluation
7. Medical condition or medication putting at undue risk
8. Medical condition that is unstable at the time of the study or that may interfere with the study
9. History of organ transplant
10. Pigmentation on the back is difficult to evaluate due to excessive hair or presence of a tattoo

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Lowest mean fluence inducing visible pigmentation | 7 days
  Lowest mean fluence inducing visible pigmentation 7 days after visible light exposure for skin where a topical antioxidant was applied compared to skin where control was applied.

SECONDARY OUTCOMES:
Mean difference in pigmentation intensity | 7 days
  Difference in pigmentation intensity between skin with antioxidant and skin with control.
Protection factor of antioxidant preparation against visible light | 7 days
  Protection factor of antioxidant preparation against visible light between antioxidant and control.
Safety of the antioxidant preparation | 7 days
  Safety of the antioxidant preparation measured by the number of adverse events and the severity of adverse events compared to control

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, FRCPC, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research Inc, Montreal, Quebec, Canada

REFERENCES:
- [Background] Mahmoud BH, Ruvolo E, Hexsel CL, Liu Y, Owen MR, Kollias N, Lim HW, Hamzavi IH. Impact of long-wavelength UVA and visible light on melanocompetent skin. J Invest Dermatol. 2010 Aug;130(8):2092-7. doi: 10.1038/jid.2010.95. Epub 2010 Apr 22. PMID 20410914
- [Background] Sklar LR, Almutawa F, Lim HW, Hamzavi I. Effects of ultraviolet radiation, visible light, and infrared radiation on erythema and pigmentation: a review. Photochem Photobiol Sci. 2013 Jan;12(1):54-64. doi: 10.1039/c2pp25152c. PMID 23111621
- [Background] Lehmann P, Schwarz T. Photodermatoses: diagnosis and treatment. Dtsch Arztebl Int. 2011 Mar;108(9):135-41. doi: 10.3238/arztebl.2011.0135. Epub 2011 Mar 4. PMID 21442060
- [Background] Terezakis NK, Bazzano GS. Retinoids: compounds important to hair growth. Clin Dermatol. 1988 Oct-Dec;6(4):129-31. doi: 10.1016/0738-081x(88)90077-6. PMID 3063367
- [Background] Porges SB, Kaidbey KH, Grove GL. Quantification of visible light-induced melanogenesis in human skin. Photodermatol. 1988 Oct;5(5):197-200. PMID 3222167
- [Background] Pandya AG, Guevara IL. Disorders of hyperpigmentation. Dermatol Clin. 2000 Jan;18(1):91-8, ix. doi: 10.1016/s0733-8635(05)70150-9. PMID 10626115
- [Background] Liebel F, Kaur S, Ruvolo E, Kollias N, Southall MD. Irradiation of skin with visible light induces reactive oxygen species and matrix-degrading enzymes. J Invest Dermatol. 2012 Jul;132(7):1901-7. doi: 10.1038/jid.2011.476. Epub 2012 Feb 9. PMID 22318388
- [Background] Ball Arefiev KL, Hantash BM. Advances in the treatment of melasma: a review of the recent literature. Dermatol Surg. 2012 Jul;38(7 Pt 1):971-84. doi: 10.1111/j.1524-4725.2012.02435.x. Epub 2012 May 14. PMID 22583339
- [Background] Chen L, Hu JY, Wang SQ. The role of antioxidants in photoprotection: a critical review. J Am Acad Dermatol. 2012 Nov;67(5):1013-24. doi: 10.1016/j.jaad.2012.02.009. Epub 2012 Mar 9. PMID 22406231
- [Background] Sheth VM, Pandya AG. Melasma: a comprehensive update: part I. J Am Acad Dermatol. 2011 Oct;65(4):689-697. doi: 10.1016/j.jaad.2010.12.046. PMID 21920241
- [Background] Kameyama K, Sakai C, Kondoh S, Yonemoto K, Nishiyama S, Tagawa M, Murata T, Ohnuma T, Quigley J, Dorsky A, Bucks D, Blanock K. Inhibitory effect of magnesium L-ascorbyl-2-phosphate (VC-PMG) on melanogenesis in vitro and in vivo. J Am Acad Dermatol. 1996 Jan;34(1):29-33. doi: 10.1016/s0190-9622(96)90830-0. PMID 8543691
- [Background] Ertam I, Mutlu B, Unal I, Alper S, Kivcak B, Ozer O. Efficiency of ellagic acid and arbutin in melasma: a randomized, prospective, open-label study. J Dermatol. 2008 Sep;35(9):570-4. doi: 10.1111/j.1346-8138.2008.00522.x. PMID 18837701
- [Background] Hwang SW, Oh DJ, Lee D, Kim JW, Park SW. Clinical efficacy of 25% L-ascorbic acid (C'ensil) in the treatment of melasma. J Cutan Med Surg. 2009 Mar-Apr;13(2):74-81. doi: 10.2310/7750.2008.07092. PMID 19298775
- [Background] Stella A, Golin R, Zanchetti A. Effects of reversible renal denervation on haemodynamic and excretory functions of the ipsilateral and contralateral kidney in the cat. J Hypertens. 1986 Apr;4(2):181-8. doi: 10.1097/00004872-198604000-00007. PMID 3519762
- [Background] Wu Y, Matsui MS, Chen JZ, Jin X, Shu CM, Jin GY, Dong GH, Wang YK, Gao XH, Chen HD, Li YH. Antioxidants add protection to a broad-spectrum sunscreen. Clin Exp Dermatol. 2011 Mar;36(2):178-87. doi: 10.1111/j.1365-2230.2010.03916.x. Epub 2010 Aug 27. PMID 20804506